CLINICAL TRIAL: NCT00799266
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled Efficacy and Safety Trial of Intravenous Zoledronic Acid Twice Yearly Compared to Placebo in Osteoporotic Children Treated With Glucocorticoids.
Brief Title: An Efficacy and Safety Trial of Intravenous Zoledronic Acid Twice Yearly in Osteoporotic Children Treated With Glucocorticoids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446H2337; 2008-001252-52 (EudraCT Number)
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, children and adolescents, zoledronic acid, chronic inflammation, Duchenne muscular dystrophy, glucocorticoids, chronic inflammatory conditions
MeSH Terms: conditions — Osteoporosis; Muscular Dystrophy, Duchenne | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Zoledronic acid (Experimental): Twice yearly 0.05 mg/kg (max 5 mg) i.v infusion (at least 30 minutes) of zoledronic acid
  Interventions: Drug: Zoledronic acid
- Placebo (Placebo Comparator): Twice yearly i.v of infusion of Placebo (similar dosing as active drug)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic acid — intravenous infusion
  Arms: Zoledronic acid
Drug: Placebo — intravenous infusion
  Arms: Placebo

SUMMARY:
This study was designed to evaluate the efficacy and safety of zoledronic acid compared to placebo in osteoporotic children treated with glucocorticoids

DETAILED DESCRIPTION:
In March 2017, Novartis stopped enrollment as the study was not feasible to be conducted due to low enrollment and other recruitment challenges. Patients receiving the treatment continued to receive the treatment per protocol.

ELIGIBILITY:
Key Inclusion Criteria:

* A diagnosis of chronic rheumatologic conditions or inflammatory bowel disease or Duchenne muscular dystrophy requiring systemic glucocorticoids (i.v. or oral) within 12 months prior to screening
* Lumbar Spine BMDZ-score of -0.5 or worse
* Evidence of at least at least 1 vertebral compression fracture of Genant Grade 1 or higher (or radiographic signs of vertebral fracture) within 1 month from Screening visit OR One or more, low-trauma, lower extremity long-bone fracture which occurred sometime within the 2 years PRECEDING enrollment in the study OR Two or more, low-trauma, upper extremity long-bone fractures which occurred sometime within the 2 years PRECEDING enrollment in the study
* Consent/assent to study participation

Key Exclusion Criteria:

* History of primary bone disease (OI, Idiopathic Juvenile Osteoporosis, Rickets/Osteomalacia)
* Any medical condition that might have interfered with the evaluation of lumbar spine BMD, such as severe scoliosis or spinal fusion. Patients with less than 3 evaluable vertebrae by Dual Energy X-ray Absorptiometry (DXA) evaluation in the region of interest lumbar 1 (L1) to lumbar 4 (L4),
* Hypocalcemia and hypophosphatemia
* Serum 25-hydroxy vitamin D concentrations of <20 ng/mL or <50 nmol/L
* estimated glomerular filtration rate (GFR) <60 mL/min/1.73 m2
* serum creatinine increase between Visit 1 and Visit 2 >0.5 mg/dL (44.2 μmol/L)
* Uncontrolled symptoms of cardiac failure or arrhythmia
* Any prior use of bisphosphonates, or high dose sodium fluoride

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2008-12-04 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Budapest, Hungary
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Soweto, Gauteng, South Africa
- United Kingdom (2):
  - Novartis Investigative Site, West Midlands, Birmingham
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Ward LM, Choudhury A, Alos N, Cabral DA, Rodd C, Sbrocchi AM, Taback S, Padidela R, Shaw NJ, Hosszu E, Kostik M, Alexeeva E, Thandrayen K, Shenouda N, Jaremko JL, Sunkara G, Sayyed S, Aftring RP, Munns CF. Zoledronic Acid vs Placebo in Pediatric Glucocorticoid-induced Osteoporosis: A Randomized, Double-blind, Phase 3 Trial. J Clin Endocrinol Metab. 2021 Nov 19;106(12):e5222-e5235. doi: 10.1210/clinem/dgab458. PMID 34228102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 12 centers in 6 countries: Australia (1), Canada (5), Hungary (1), United Kingdom (2), Russian Federation (2), and South Africa (1).
Pre-assignment Details: The Participant Flow and Baseline Characteristics were done on the Intention-to-treat (ITT) population. All efficacy analyses were done on the Modified Intention-to-treat (MITT) population and all safety analyses were based on Safety population.
Period: Overall Study
Arm/Group | Zoledronic Acid | Placebo
Started (All randomized patients (ITT)) | 18 | 16
Modified Intention-to-treat (MITT) (All patients with baseline and at least one post-baseline lumbar spine BMD Z-score) | 17 | 16
Safety Set (All patients with at least one infusion of study drug) | 18 | 16
Completed | 15 | 15
Not Completed | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Subject withdrew consent | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Participant Flow and Demographics (age/gender/race) were done on the Intention-to-treat (IIT) population whereas the Baseline disease characteristics were on the Modified Intention-to-treat (MITT). All efficacy analyses were done on the Modified Intention-to-treat (MITT) population and all safety analyses were based on Safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Placebo | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.0 (3.50) | 12.3 (3.42) | 12.6 (3.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 13 | 14 | 27
  Black | 2 | 1 | 3
  Asian | 2 | 0 | 2
  Native American | 1 | 1 | 2
  Pacific Islander | 0 | 0 | 0
  Othe | 0 | 0 | 0
Lumbar Spine Bone Mineral Density (BMD) Z-score [Mean (Standard Deviation); unit: Z-score] — Lumbar Spine Bone Mineral Density (BMD) Z-score in the Modified Intention-to-treat (MITT) population. No imputation done at Baseline. Bone mass, as measured by DXA, is reported as BMC (g) or areal BMD (g/cm2). These values are compared with reference values from healthy youth of similar age, sex, and race/ ethnicity to calculate a z score, the number of SDs from the expected mean. A BMC or BMD z score that is >2 SDs below expected (< -2.0) is referred to as "low for age". Population: Modified Intention-to-treat (MITT) population = All patients with baseline and at least one post-baseline lumbar spine BMD Z-score
  Z-score
    number analyzed (Participants) | 17 | 16 | 33
    (all) | -2.127 (0.7863) | -2.379 (0.8975) | -2.249 (0.8385)
Lumbar Spine Bone Mineral Content (BMC) [Mean (Standard Deviation); unit: gram (g)] — Lumbar Spine Bone Mineral Content (BMC) in the Modified Intention-to-treat (MITT) population. No imputation done at Baseline. Population: Modified Intention-to-treat (MITT) population = All patients with baseline and at least one post-baseline lumbar spine BMD Z-score
  gram (g)
    number analyzed (Participants) | 17 | 16 | 33
    (all) | 31.886 (15.1062) | 22.605 (6.6054) | 27.386 (12.5195)
Total body Bone Mineral Content (BMC) [Mean (Standard Deviation); unit: gram (g)] — Total body Bone Mineral Content (BMC) in the Modified Intention-to-treat (MITT) population. No imputation done at Baseline. Population: Modified Intention-to-treat (MITT) population = All patients with baseline and at least one post-baseline lumbar spine BMD Z-score
  gram (g)
    number analyzed (Participants) | 16 | 14 | 30
    (all) | 1550.556 (592.0670) | 1050.610 (253.0759) | 1317.248 (523.8133)
Serum Procollagen type 1 amino-terminal propeptide (P1NP) [Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)] — Serum Procollagen type 1 amino-terminal propeptide (P1NP) in the Modified Intention-to-treat (MITT) population. No imputation done at Baseline. Population: Modified Intention-to-treat (MITT) population = All patients with baseline and at least one post-baseline lumbar spine BMD Z-score
  nanogram per milliliter (ng/mL)
    number analyzed (Participants) | 16 | 14 | 30
    (all) | 313.54 (284.541) | 368.90 (235.226) | 339.37 (259.750)
Serum Bone specific alkaline phosphatase (BSAP) [Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)] — Serum Bone specific alkaline phosphatase (BSAP) in the Modified Intention-to-treat (MITT) population. No imputation done at Baseline. Population: Modified Intention-to-treat (MITT) population = All patients with baseline and at least one post-baseline lumbar spine BMD Z-score
  nanogram per milliliter (ng/mL)
    number analyzed (Participants) | 16 | 14 | 30
    (all) | 31.559 (22.6619) | 43.414 (32.8200) | 37.092 (28.0122)
Serum Cross linked N-telopeptide (NTX) [Mean (Standard Deviation); unit: nmol BCE/L] — Serum Cross linked N-telopeptide (NTX) in the Modified Intention-to-treat (MITT) population. No imputation done at Baseline. Population: Modified Intention-to-treat (MITT) population = All patients with baseline and at least one post-baseline lumbar spine BMD Z-score
  nmol BCE/L
    number analyzed (Participants) | 16 | 14 | 30
    (all) | 34.359 (22.0490) | 39.192 (14.5823) | 36.615 (18.7829)
Serum Tartrate-resistant acid phosphatase isoform 5b (TRAP-5b) [Mean (Standard Deviation); unit: U/L] — Serum Tartrate-resistant acid phosphatase isoform 5b (TRAP-5b) in the Modified Intention-to-treat (MITT) population. No imputation done at Baseline. Population: Modified Intention-to-treat (MITT) population = All patients with baseline and at least one post-baseline lumbar spine BMD Z-score
  U/L
    number analyzed (Participants) | 16 | 14 | 30
    (all) | 7.010 (2.9998) | 8.595 (4.5650) | 7.750 (3.8266)
Vertebral Morphometry (mid-to-posterior height ratio) [Mean (Standard Deviation); unit: mid-to-posterior height ratio] — Vertebral Morphometry (mid-to-posterior height ratio) in the Modified Intention-to-treat (MITT) population. Calculation was done using average ratio between mid-height and posterior height from L1 to L4 and analysis of covariance model was used with treatment, pooled centers, underlying condition treated with glucocordicoids and baseline value as explanatory variables and pooled centers as random effect. Population: Modified Intention-to-treat (MITT) population = All patients with baseline and at least one post-baseline lumbar spine BMD Z-score
  mid-to-posterior height ratio
    number analyzed (Participants) | 10 | 13 | 23
    (all) | 0.982 (0.0428) | 0.976 (0.0788) | 0.979 (0.0643)
Second metacarpal cortical width [Mean (Standard Deviation); unit: millimeter (mm)] — Second metacarpal cortical width in the Modified Intention-to-treat (MITT) population. Metacarpal cortical width of "0" was not included. An analysis of covariance model used with treatment, pooled centers, underlying condition treated with glucocorticoids at baseline value as explanatory variables and pooled centers as random effect. Population: Modified Intention-to-treat (MITT) population = All patients with baseline and at least one post-baseline lumbar spine BMD Z-score
  millimeter (mm)
    number analyzed (Participants) | 9 | 12 | 21
    (all) | 0.40 (0.194) | 0.41 (0.144) | 0.40 (0.163)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) Z-score at Month 12
Description: Lumbar Spine Bone Mineral Density (BMD) Z-score was determined by the central imaging vendor before first treatment and at Month 12. The methods to be used to measure Lumbar Spine BMD Z-score were described in the respective DXA Manuals provided by central imaging vendor. Positive changes from baseline indicated an improvement in condition.
Time Frame: Month 12
Population: The Modified Intention-to-treat (MITT) population, which consisted of all randomized patients who had both baseline and at least one post-baseline lumbar spine BMD Z-score, was considered.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
Z-score | 0.582 (0.1279) | 0.168 (0.1449)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Lumbar Spine BMD Z-score at Month 12; Test type: Superiority — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.0392, ANCOVA; Difference in LS mean = 0.414, 95% CI 2-sided [0.022 to 0.806]

2. Secondary Outcome: Mean Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) Z-score at Month 6
Description: Lumbar Spine Bone Mineral Density (BMD) Z-score was determined by the central imaging vendor before first treatment and at Month 6. The methods to be used to measure Lumbar Spine BMD Z-score were described in the respective DXA Manuals provided by central imaging vendor. Positive changes from baseline indicated an improvement in condition.
Time Frame: Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
Z-score | 0.447 (0.13) | 0.157 (0.14)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Lumbar Spine BMD Z-score at Month 6; Test type: Superiority — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.1322, ANCOVA; Difference in LS mean = 0.290, 95% CI 2-sided [-0.094 to 0.673]

3. Secondary Outcome: Mean Change From Baseline in Lumbar Spine BMC at Month 6 and 12
Description: Lumbar Spine BMC was determined by the central imaging vendor before first treatment and at Months 6 and 12. The methods to be used to measure BMC were described in the respective DXA Manuals.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
g
  Lumbar Spine (LS) BMC Change at Month 6: number analyzed (Participants) | 16 | 15
  Lumbar Spine (LS) BMC Change at Month 6 | 4.110 (0.63) | 2.131 (0.70)
  Lumbar Spine (LS) BMC Change at Month 12: number analyzed (Participants) | 16 | 15
  Lumbar Spine (LS) BMC Change at Month 12 | 6.450 (1.18) | 4.295 (1.32)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Lumbar Spine BMC at Month 6; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.0409, ANCOVA; Difference in LS mean = 1.979, 95% CI 2-sided [0.089 to 3.869]
Statistical Analysis 2: Comparison: Zoledronic Acid vs Placebo; Lumbar Spine BMC at Month 12; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.2340, ANCOVA; Difference in LS mean = 2.155, 95% CI 2-sided [-1.488 to 5.798]

4. Secondary Outcome: Mean Change From Baseline in Total Body BMC at Month 6 and 12
Description: Total body BMC was all determined by the central imaging vendor before first treatment and at Months 6 and 12. The methods to be used to measure BMC were described in the respective DXA Manuals.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
g
  Total BMC Change at Month 6: number analyzed (Participants) | 15 | 13
  Total BMC Change at Month 6 | 129.272 (24.23) | 95.214 (28.74)
  Total BMC Change at Month 12: number analyzed (Participants) | 15 | 12
  Total BMC Change at Month 12 | 220.805 (42.74) | 140.064 (51.90)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Total Body BMC at Month 6; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.3827, ANCOVA; Difference in LS mean = 34.058, 95% CI 2-sided [-45.385 to 113.502]
Statistical Analysis 2: Comparison: Zoledronic Acid vs Placebo; Total Body BMC at Month 12; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.2634, ANCOVA; Difference in LS mean = 80.741, 95% CI 2-sided [-65.602 to 227.084]

5. Secondary Outcome: Mean Change From Baseline in Serum P1NP at Months 6 and 12
Description: Serum Procollagen type 1 amino-terminal propeptide (P1NP) was collected before first treatment (baseline) and at Months 6 and Month 12 according to the instructions provided in the Laboratory Manual. The samples were analyzed in batches at the laboratory.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nanogram per milliliter (ng/mL)
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
nanogram per milliliter (ng/mL)
  P1NP Change at Month 6: number analyzed (Participants) | 14 | 15
  P1NP Change at Month 6 | -134.285 (48.80) | 77.497 (56.15)
  P1NP Change at Month 12: number analyzed (Participants) | 15 | 15
  P1NP Change at Month 12 | -230.966 (59.1977) | 150.166 (68.0933)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Serum P1NP at Month 6; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.0631, ANCOVA; Difference in LS mean = -211.782, 95% CI 2-sided [-363.765 to -59.800]
Statistical Analysis 2: Comparison: Zoledronic Acid vs Placebo; Serum P1NP at Month 12; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.0049, ANCOVA; Difference in LS mean = -381.132, 95% CI 2-sided [-565.416 to -196.848]

6. Secondary Outcome: Mean Change From Baseline in BSAP at Months 6 and 12
Description: Bone specific alkaline phosphatase (BSAP) were collected before first treatment (baseline) and at Months 6 and Month 12 according to the instructions provided in the Laboratory Manual. The samples were analyzed in batches at the laboratory.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nanogram per milliliter (ng/mL)
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
nanogram per milliliter (ng/mL)
  BSAP Change at Month 6: number analyzed (Participants) | 14 | 15
  BSAP Change at Month 6 | -7.413 (3.63) | 3.810 (4.05)
  BSAP Change at Month 12: number analyzed (Participants) | 15 | 15
  BSAP Change at Month 12 | -13.984 (4.3814) | 6.450 (4.9010)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Serum BSAP at Month 6; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.2129, ANCOVA; Difference in LS mean = -11.223, 95% CI 2-sided [-22.595 to 0.149]
Statistical Analysis 2: Comparison: Zoledronic Acid vs Placebo; Serum BSAP at Month 12; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.0215, ANCOVA; Difference in LS mean = -20.435, 95% CI 2-sided [-33.960 to -6.909]

7. Secondary Outcome: Mean Change From Baseline in Serum NTX at Months 6 and 12
Description: Serum Cross linked N-telopeptide (NTX) were collected before first treatment (baseline) and at Months 6 and Month 12 according to the instructions provided in the Laboratory Manual. The samples were analyzed in batches at the laboratory.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol BCE/L
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
nmol BCE/L
  NTX Change at Month 6: number analyzed (Participants) | 14 | 15
  NTX Change at Month 6 | -13.746 (4.23) | 7.192 (4.74)
  NTX Change at Month 12: number analyzed (Participants) | 15 | 15
  NTX Change at Month 12 | -20.134 (3.76) | 7.440 (4.23)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Serum NTX at Month 6; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.0254, ANCOVA; Difference in LS mean = -20.938, 95% CI 2-sided [-33.766 to -8.110]
Statistical Analysis 2: Comparison: Zoledronic Acid vs Placebo; Serum NTX at Month 12; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.0002, ANCOVA; Difference in LS mean = -27.574, 95% CI 2-sided [-39.037 to -16.111]

8. Secondary Outcome: Mean Change From Baseline in Serum TRAP-5b at Months 6 and 12
Description: Serum Tartrate-resistant acid phosphatase isoform 5b (TRAP 5b) was collected before first treatment (baseline) and at Months 6 and Month 12 according to the instructions provided in the Laboratory Manual. The samples were analyzed in batches at the laboratory.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
U/L
  TRAP 5b Change at Month 6: number analyzed (Participants) | 14 | 15
  TRAP 5b Change at Month 6 | -1.561 (0.65) | 0.313 (0.74)
  TRAP 5b Change at Month 12: number analyzed (Participants) | 14 | 15
  TRAP 5b Change at Month 12 | -1.728 (0.73) | 0.109 (0.81)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Serum TRAP-5b at Month 6; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.2178, ANCOVA; Difference in LS mean = -1.874, 95% CI 2-sided [-3.931 to 0.182]
Statistical Analysis 2: Comparison: Zoledronic Acid vs Placebo; Serum TRAP-5b at Month 12; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.1840, ANCOVA; Difference in LS mean = -1.837, 95% CI 2-sided [-4.103 to 0.429]

9. Secondary Outcome: Number of Participants With New Vertebral Fractures at Month 12
Description: New vertebral fractures were defined as fractures of Genant Grade 1 or higher that occurred at lumbar or thoracic spine from first dose infusion to the end of the study.
Time Frame: Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
Participants | 0 | 2
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; New vertebral fractures at Month 12; Test type: Other — The number and percentage of patients with new vertebral fractures at Month 12 were presented by treatment group and between-treatment differences were evaluated using Fisher's exact test; p = 0.2258, Fisher Exact

10. Secondary Outcome: Mean Change From Baseline in Vertebral Morphometry at Month 12
Description: Vertebral morphometry (or concave index) was calculated using the average ratio between mid-height and posterior height from L1 to L4 and performed by a central reader.
Time Frame: Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
Ratio | -0.018 (0.01) | -0.0003 (0.01)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Vertebral morphometry at Month 12; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.3180, ANCOVA; Difference in LS mean = -0.018, 95% CI 2-sided [-0.055 to 0.019]

11. Secondary Outcome: Percentage of Patients With Reduction in Pain at Months 3, 6, 9 and 12
Description: Pain was evaluated at each visit (in office and telephone visit) at randomization, Months 3, 6, 9 and 12 using the Faces Pain Scale-Revised (FPS-R). Children were selecting the face that best fits their pain. The pain score ranged from 0 (No Pain) to 10 (Very Much Pain). The reduction in pain from baseline by visit was evaluated based on whether or not patients had a decrease in their FPS-R from baseline. If pain remained the same or worsened from baseline a patient was classified as '0' and if the pain scale decreased then the patient was classified as '1'.
Time Frame: Month 3, Month 6, Month 9 and Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
Percentage of Patients
  Month 3: number analyzed (Participants) | 16 | 13
  Month 3 | 37.5 | 53.8
  Month 6: number analyzed (Participants) | 16 | 14
  Month 6 | 37.5 | 50.0
  Month 9: number analyzed (Participants) | 15 | 13
  Month 9 | 33.3 | 46.2
  Month 12: number analyzed (Participants) | 16 | 14
  Month 12 | 31.3 | 57.1
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Reduction in Pain at Month 3; Test type: Other — Presented by treatment group and evaluated using a logistic regression model with treatment, pooled centers, underlying condition treated with glucocorticoids and baseline pain score as explanatory variables; p = 0.5226, Regression, Logistic; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.04 to 5.20]
Statistical Analysis 2: Comparison: Zoledronic Acid vs Placebo; Reduction in Pain at Month 6; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.5220, Regression, Logistic — >999.99 (<0.01, >999.99); Odds Ratio (OR) = 999.99, 95% CI 2-sided [0.01 to 999.99]
Statistical Analysis 3: Comparison: Zoledronic Acid vs Placebo; Reduction in Pain at Month 9; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.6019, Regression, Logistic; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.04 to 6.22]
Statistical Analysis 4: Comparison: Zoledronic Acid vs Placebo; Reduction in Pain at Month 12; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.9652, Regression, Logistic — 0.45 (<0.01, >999.99); Odds Ratio (OR) = 0.45, 0.9652% CI 2-sided [0.01 to 999.99]

12. Secondary Outcome: Mean Change From Baseline in 2nd Metacarpal Cortical Width at Month 12
Description: Left posteroanterior (PA) hand/wrist X-ray were taken at Visit 1 and at the Month 12 visit to assess bone age and the between-treatment differences for change in 2nd metacarpal cortical width at Month 12 relative to baseline. If a fracture of the left upper extremity precluded radiographic imaging, then the right hand was evaluated for this purpose. In this case, the right hand was be imaged at both Visit 1 and at Month 12. The information was used in the assessment of bone density.
Time Frame: Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 17 | 16
millimeter (mm) | -0.01 (0.040) | 0.03 (0.047)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; 2nd metacarpal cortical width at Month 12; Test type: Other — Difference in least squares (LS) = LS mean for the zoledronic acid group-LS mean for the placebo group; p = 0.5165, ANCOVA; Difference in LS mean = -0.04, 95% CI 2-sided [-0.17 to 0.09]

13. Secondary Outcome: Urinary Concentration of Zoledronic Acid at Month 12
Description: Urine was collected overnight or for at least 4 waking hours from all patients able to provide specimens, to measure urinary concentration of zoledronic acid at Month 12. Only descriptive analysis done.
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 17
ng/mL | 1643.3 (2846.34)

14. Secondary Outcome: Safety of Zoledronic Acid for the Treatment of Osteoporotic Children Treated With Glucocorticoids
Description: Analysis of absolute and relative frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC) to demonstrate that zoledronic acid is safe for the treatment of osteoporotic children treated with glucocorticoids through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive analysis done.
Time Frame: Baseline through Month 12
Population: The Safety population, which consisted of all patients who had been exposed to at least one infusion of study drug, was considered.
Measure: Number; unit: Percentage of Participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 18 | 16
Percentage of Participants
  AEs by Primary System Organ Class (SOC): number analyzed (Participants) | 15 | 12
  AEs by Primary System Organ Class (SOC) | 83.3 | 75.0
  SAEs by Primary System Organ Class (SOC): number analyzed (Participants) | 5 | 1
  SAEs by Primary System Organ Class (SOC) | 27.8 | 6.3
  Deaths by Primary System Organ Class (SOC): number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 9 years and 3 months.
Arm/Group | Zoledronic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 5/18 | 1/16
Other Adverse Events (participants affected / at risk) | 14/18 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=18) | Placebo (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Acute phase reaction (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=18) | Placebo (N=16)
Tachycardia (Cardiac disorders) | 3 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 0
Dry eye (Eye disorders) | 0 | 1
Eye disorder (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Tooth erosion (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Acute phase reaction (General disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
Pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 3 | 1
Thirst (General disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood iron decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Lethargy (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Sleep talking (Psychiatric disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 | 0
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-10-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT00799266/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT00799266/SAP_001.pdf